CLINICAL TRIAL: NCT01142037
Title: Development of a Biomarker for Dietary Furanocoumarins
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2009NTLS107; 0909M72358 (Other: IRB, University of Minnesota); 1K07CA128952-01A2 (NIH)
Record Dates: First submitted 2010-06-09; First posted 2010-06-11 (Estimated); Last update posted 2014-08-22 (Estimated); Status verified 2014-08

CONDITIONS: Cancer; Healthy
Keywords: Healthy volunteer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Furanocoumarin (Experimental): Includes participants first refraining from eating foods with furanocoumarins for one week, followed by 2 weeks of increasing furanocoumarin consumption. Participants will be asked to consume cooked parsnips and parsley.
  Interventions: Dietary Supplement: Cooked parsnips with parsley

INTERVENTIONS:
Dietary Supplement: Cooked parsnips with parsley — Beginning on Day 9 participants will be given cooked parsnips with parsley at a dose of 2 grams total apiaceous vegetable/kilogram body weight for period 1, and 4 gram/kilogram body weight for period 2.

SUMMARY:
Certain plant foods are high in furanocoumarins. Test tube and animal studies suggest that furanocoumarins may help prevent cancer. It is difficult to determine in humans if furanocoumarins do prevent cancer because there isn't an objective way to tell who has eaten these compounds. This study will develop a urine test to determine if an individual ate foods that contain furanocoumarins.

ELIGIBILITY:
Inclusion Criteria:

* Must be at least 18 years of age
* Healthy

Exclusion Criteria:

* History of gastrointestinal, hepatic or renal disorder
* Currently taking any prescription or over-the-counter medication
* Currently taking any herbal supplement
* Pregnant or lactating
* Allergies to foods that will be used (parsnips and parsley)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-10; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Urinary Biomarker Results for Dietary Furanocoumarins | Week 1
  determine the optimal conditions for furanocoumarin identification and quantification in human urine

SECONDARY OUTCOMES:
Mean Concentration of Dietary Furanocoumarin in Urine | Week 1, 2 and 3
  Determine dose response of dietary furanocoumarin in urine - Comparison of Pre-Dose, Low-Dose and High Dose diet of furanocoumarin in subjects' urine collected (ng/ml).

CONTACTS AND LOCATIONS:
Overall Officials: Sabrina Peterson, Ph.D., Principal Investigator — University of Minnesota
Locations (1):
- Department of Food Science and Nutrition, University of Minnesota, Saint Paul, Minnesota, United States